CLINICAL TRIAL: NCT01806142
Title: Effects of Medium-Chain Triglycerides on Chylomicron Secretion and Expression of Genes That Regulate Intestinal Lipid Metabolism in Men With Dyslipidemia Associated With the Metabolic Syndrome
Acronym: MCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Patrick Couture, MD, FRCP, PhD, Laval University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: INAF-C10-08-053
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome | interventions — Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medium-chain triglycerides (Experimental): During Medium-Chain Triglycerides (MCT period), participant will asked to consume two pastries per day that will provide a total of 20 g of MCT/day for 4 weeks.
  Interventions: Other: Medium-chain triglycerides
- Corn oil (Active Comparator): During Corn oil period (Control period), participant will asked to consume two pastries per day that will provide a total of 20 g of corn oil/day for 4 weeks.
  Interventions: Other: Corn oil

INTERVENTIONS:
Other: Medium-chain triglycerides — During Medium-Chain Triglycerides (MCT period), participant will asked to consume two pastries per day that will provide a total of 20 g of MCT/day for 4 weeks.
  Arms: Medium-chain triglycerides
Other: Corn oil — During Corn oil period (Control period), participant will asked to consume two pastries per day that will provide a total of 20 g of corn oil/day for 4 weeks.
  Arms: Corn oil

SUMMARY:
Several lines of evidence indicate that a significant proportion of cardiovascular disease (CVD) events are attributable to the presence of a cluster of metabolic abnormalities and perturbations, defined as the metabolic syndrome. It has been estimated that approximately 25% of the North American adult population is living with the metabolic syndrome. Recent studies from the investigators group show that overaccumulation of atherogenic triglyceride-rich lipoproteins (TRL) seen in insulin-resistant patients is partly due to increased production rate of intestinally derived apolipoprotein (apo) B-48-containing lipoproteins. This is of interest because substantial evidence exists indicating that elevated levels of intestinal lipoproteins are associated with increased CVD risk. In this regard, there is some evidence that medium-chain triglycerides (MCTs) may beneficially modify lipoprotein metabolism in hypertriglyceridemic patients. However, as emphasized in the body of this grant proposal, the specific impact of MCTs on the intestinal lipoprotein secretion and on expression of genes that regulate intestinal lipid absorption and chylomicron synthesis has not yet been investigated in humans.

The general objective of the proposed research is to investigate the mechanisms by which MCTs beneficially modify intestinal lipoprotein metabolism in patients with the metabolic syndrome. The primary hypothesis is that MCT supplementation will decrease plasma levels of intestinal lipoproteins by reducing secretion of these particles.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18-60 years
* Waist circumference > 102 cm
* HDL-cholesterol < 1.1 mmol/L
* Triglycerides > 1.7 mmol/L
* Fasting blood glucose > 6.1 mmol/L
* Normal blood pressure (<130/85)

Exclusion Criteria:

* Women
* Men < 18 or > 60 years
* Smokers (> 1 cigarette/day)
* Body weight variation > 10% during the last 6 months prior to the study baseline
* Subjects with a previous history of cardiovascular disease
* Subjects with type 2 diabetes
* Subjects with a monogenic dyslipidemia
* Subjects on hypertension medications or medications known to affect lipoprotein metabolism or the integrity of gastrointestinal mucosa
* Subjects with endocrine or gastrointestinal disorders
* History of alcohol or drug abuse within the past 2 years
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in TRL apolipoprotein B48 (apoB-48) production rate. | At week 4 and week 10 (at the end of the two 4-weeks supplementation).

SECONDARY OUTCOMES:
Changes in duodenal expression of genes that regulate intestinal lipid absorption. | At week 4 and week 10 (at the end of the two 4-weeks supplementation).
  Genes that regulate intestinal lipid absorption that will be measured are Niemann-Pick C1-like 1 (NPC1L1), Adenosine triphosphate(ATP)-binding cassette transporters (ABCG5/8), Fatty Acid Binding Protein (FABP), Sterol Regulatory Element Binding Protein (SREBP-1c).
Changes in duodenal expression of genes that regulate intestinal lipid synthesis. | At week 4 and week 10 (at the end of the two 4-weeks supplementation).
  Genes that regulate intestinal lipid synthesis that will be measured are Acyl-Coenzyme A(CoA):diacylglycerol acyltransferase (DGAT), Acyl-CoA:cholesterol O-acyltransferase 2 (ACAT2) and 3-hydroxy-methylglutaryl-CoA reductase (HMG CoA reductase).
Change in synthesis of apoB-48 containing lipoproteins (Microsomal triglyceride transfer protein (MTP), apoB-48). | At week 4 and week 10 (at the end of the two 4-weeks supplementation).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD,FRCP,PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada

REFERENCES:
- [Derived] Tremblay AJ, Lamarche B, Labonte ME, Lepine MC, Lemelin V, Couture P. Dietary medium-chain triglyceride supplementation has no effect on apolipoprotein B-48 and apolipoprotein B-100 kinetics in insulin-resistant men. Am J Clin Nutr. 2014 Jan;99(1):54-61. doi: 10.3945/ajcn.113.068767. Epub 2013 Oct 30. PMID 24172309